CLINICAL TRIAL: NCT06707545
Title: In Situ Analysis of the Optical Quality and Visual Solvency of Eyes Implanted Bilaterally With the Asqelio™ EDoF Toric Extended-focus Intraocular Lens
Brief Title: Visual Quality and Performance of Eyes With Asqelio™ EDoF Toric Lenses
Status: Completed | Type: Observational
Sponsor: AST Products, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ASQE022022
Record Dates: First submitted 2024-11-24; First posted 2024-11-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2024-11

CONDITIONS: Cataract; Presbyopia Correction
Keywords: intraocular lens; extended depth-of-focus; cataract surgery; optical quality
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Asqelio EDOF: Patients submitted to cataract surgery and implanted with the extended depth-of-focus intraocular lens Asqelio EDOF Toric
- Monofocal IOL: Patients submitted to cataract surgery and implanted with the TECNIS 1-Piece monofocal intraocular lens

SUMMARY:
This study evaluates the optical quality and clinical performance of the Asqelio™ EDOF Toric intraocular lens (IOL) in patients undergoing cataract surgery or refractive lensectomy. The Asqelio™ EDOF Toric IOL aims to provide improved vision at various distances and correct astigmatism compared to monofocal IOLs. Postoperative outcomes, including visual clarity, refractive correction, and patient satisfaction, will be assessed three months after surgery.

DETAILED DESCRIPTION:
Cataract surgery is one of the most common procedures worldwide, typically involving the replacement of the cloudy natural lens with an intraocular lens (IOL). Traditional monofocal IOLs correct vision for a single distance but do not address intermediate or near vision, leading to dependence on glasses. The Asqelio™ EDOF Toric IOL is designed to provide extended depth of focus, smoother transitions across distances, and astigmatism correction, potentially enhancing overall visual quality and reducing the need for glasses.

This study compares the optical performance and patient outcomes of the Asqelio™ EDOF Toric IOL with those of monofocal IOLs. Key measures include optical quality, visual acuity at multiple distances, refractive correction, and patient-reported satisfaction. Results will be collected during a three-month postoperative follow-up. The findings aim to inform the effectiveness of the Asqelio™ EDOF Toric IOL in improving visual outcomes and quality of life for patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 50 years or older who have undergone cataract surgery with phacoemulsification or refractive lensectomy, with bilateral implantation of the Asqelio EDOF toric IOL model ETLIO130C/ETPIO130C with a cylinder value of 0.0 D, or the spherical monofocal J&J TECNIS 1-Piece IOL model ZCB00.
* Patients who have signed the informed consent form.
* Clear intraocular media, except for the presence of cataracts in both eyes prior to surgery.
* Postoperative potential visual acuity of 20/25 or better

Exclusion Criteria:

* Preoperative corneal astigmatism greater than 1.00D.
* Patients who do not provide informed consent.
* Patients who do not understand the study procedure.
* Previous corneal surgery or trauma.
* Irregular cornea (e.g., keratoconus).
* Choroidal hemorrhage.
* Microphthalmos.
* Severe corneal dystrophy.
* Uncontrolled or medically controlled glaucoma.
* Clinically significant macular changes.
* Severe concomitant ocular disease.
* Cataract unrelated to aging.
* Severe optic nerve atrophy.
* Diabetic retinopathy.
* Proliferative diabetic retinopathy.
* Amblyopia.
* Extremely shallow anterior chamber.
* Severe chronic uveitis.
* Pregnant or breastfeeding.
* Rubella.
* Mature/dense cataract preventing preoperative fundus examination.
* Previous retinal detachment.
* Concurrent participation in another drug or clinical device investigation.
* Expectation of needing another ocular surgery during the study period

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients participating in the study will have been implanted with either the spherical monofocal intraocular lens (IOL) J&J TECNIS® 1-Piece model ZCB00 (Control Group), manufactured by Johnson & Johnson Vision (Jacksonville, USA), or the extended depth of focus (EDOF) toric IOL Asqelio™ model ETLIO130C/ETPIO130C (Study Group) from AST Products, Inc., Billerica, USA, with a cylinder value of 0.0 D. All patients will be treated according to standard clinical practice, meaning that both the preoperative evaluation and the surgical procedure for IOL implantation will have been completed prior to their inclusion in the study
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-05-14 (Actual)

PRIMARY OUTCOMES:
Ocular dispersion index (OSI) | Three months after intraocular lens implantation
  OSI value represents the ratio of the amount of light within an annular area of 12 to 20 arc minute and the light corresponding to a circular area of one minute of arc around the central peak. Determined using the OQAS II double pass system
Higher order aberrations Root Mean Square (HORMS) | Three months after intraocular lens implantation
  The RMS value for higher order aberrations is calculated from the wavefront error map, determined using Hartmann-Shack wavefront aberrometry. Measured in microns
Ocular Spherical Aberration | Three months after intraocular lens implantation
  Ocular spherical aberration was determined using Hartmann-Shack wavefront aberrometry. Measured in microns.

SECONDARY OUTCOMES:
Monocular visual acuity for distance vision with correction (CDVA) | Three months after intraocular lens implantation
  The VA with its best correction placed under photopic conditions was determined monocularly at a distance of 4 meters. Measured in LogMAR units
Monocular visual acuity for distance vision without correction (UDVA) | Three months after intraocular lens implantation
  The VA without correction under photopic conditions was determined monocularly at a distance of 4 meters. Measured in LogMAR units
Monocular visual acuity for intermediate vision with correction for distance (DCIVA) | Three months after intraocular lens implantation
  The VA with its best correction placed under photopic conditions was determined monocularly at a distance of 67 centimeters. Measured in LogMAR units
Monocular visual acuity for intermediate vision without correction (UIVA) | Three months after intraocular lens implantation
  The VA without correction under photopic conditions was determined monocularly at a distance of 67 centimeters. Measured in LogMAR units
Monocular visual acuity for near vision with correction for distance (DCNVA) | Three months after intraocular lens implantation
  The VA with its best correction placed under photopic conditions was determined monocularly at a distance of 40 centimeters. Measured in LogMAR units
Monocular visual acuity for near vision without correction (UNVA) | Three months after intraocular lens implantation
  The VA without correction under photopic conditions was determined monocularly at a distance of 40 centimeters. Measured in LogMAR units
Postoperative refractive error | Three months after intraocular lens implantation
  Residual refractive error. Determined by manifest refraction. Measured in diopters
Monocular Contrast sensitivity | Three months after intraocular lens implantation
  Determined using the best-corrected Pelli-Robson test. Determined in logCS units
Binocular Contrast sensitivity | Three months after intraocular lens implantation
  Determined using the best-corrected Pelli-Robson test. Determined in logCS units
Defocus curve | Three months after intraocular lens implantation
  Binocular defocus curve obtained for the EDOF IOL group by varying the vergence of the stimulus from -4.0 D to +2.0 D in steps of 0.5 D with the best correction for distance vision
CATQuest 9SF | Three months after surgery
  Patient-reported outcomes on satisfaction and difficulty performing task after surgery. Obtained for the EDOF IOL group only. Each of the 9 items is scored using the Likert scale, from 1 for no difficulty/very satisfied, to 4 for very great difficulty/very dissatisfied, with higher scores indicating worse visual function.
Visual Symptoms questionnaire | Three months after surgery
  Questionnaire exploring the frequency, intensity and bothersome of different visual symptoms. Obtained from the subjects in the EDOF IOL group only.The scoring of these responses ranges from 0 for Never/None to 3 for Very Often/Severe/A lot, with higher scores indicating worse quality of vision

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Cano, MD, PhD, Principal Investigator — Hospital La Arruzafa
Locations (1):
- Hospital La Arruzafa, Córdoba, Cordoba, Spain

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data (IPD) for this study to ensure the confidentiality and privacy of our participants